CLINICAL TRIAL: NCT02543424
Title: Studies of the Diagnosis, Rehabilitation and Links Between Motor and Cognitive Functions in Acquired and Developmental Brain Damaged Patients
Brief Title: Motor and Cognitive Functions in Acquired and Developmental Brain Damaged Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/10FEV/053
Record Dates: First submitted 2015-08-12; First posted 2015-09-07 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Palsy; Perceptual Disorders; Hemiparesis
MeSH Terms: conditions — Cerebral Palsy; Perceptual Disorders; Paresis | interventions — Neuropsychological Tests

ARMS (2):
- Patient group (Experimental): Brain damaged adults with either hemiparesis and/or hemineglect. Brain damaged children with developmental and/or acquired disease inducing hemiparesis and/or hemineglect.
  Interventions: Behavioral: Motor, cognitive and neuropsychological assessment
- Control group (Sham Comparator): Healthy adults and children.
  Interventions: Behavioral: Motor, cognitive and neuropsychological assessment

INTERVENTIONS:
Behavioral: Motor, cognitive and neuropsychological assessment — Cognitive and motor testing and/or experimental cognitive or motor changes and/or cognitive or motor rehabilitation depending on part of the study investigated.

SUMMARY:
Neurological pathologies cause important and permanent disabilities in every day life. These pathologies can follow stoke, affecting two people per one thousand each year or cerebral palsy, affecting two births per one thousand each year. To date, the diagnosis and the rehabilitation of motor and cognitive problems has been carried out separately by different domains. For example, physiotherapists have focused on motor problems and neuropsychologists have focused on cognitive functions. However, a number of studies have demonstrated a link between motor and cognitive abilities in adults and children. The present study has three main aims: (1) to better evaluate motor and cognitive problems in brain damaged patients (all ages), (2) to understand the link between motor and cognitive abilities in patients and healthy participants and, (3) to propose new types of therapies based on the link between motor and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Congenital cerebral palsy and acquired brain injury children and adult patients
* Presenting upper limb paresis and/or hemineglect
* Between the age of 3 to 90.
* Able to understand and carry out simple verbal instruction

Exclusion Criteria:

* IQ < 70
* Severe aphasia, attentional disorder or psychiatric disorders
* Neurodegenerative disorders

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Kinematics | Change from Baseline (T0) in kinematics at an expected average of 1 week (T1), 2 months (T2) and 3 months (T3).
  Kinematics will be measured with a robotic tool called the REAplan. This tool is a distal effector robotic device that enables the patients to perform upper limb movements in a horizontal plane. The robot comprises a distal effector, a visual interface for the patient and a visual interface for the experimenter. It is fitted with incremental position sensors allowing the record of the distal effector's trajectory in the X and Y plane as function of time (125 Hz). From these records, all kind of quantitative and objective indices of upper limb quality of movement can be computed. Motor and cognitive tasks have been created on this device and have to be validated. These new tools on the robot provide a more accurate measure to better understand the participant's motor and cognitive functioning through kinematics analyses. Moreover, the robot can be used as a rehabilitative device, providing cognitive and motor assistance for specific exercises depending on participant performance.

SECONDARY OUTCOMES:
Standardized cognitive and motor assessment | Change from Baseline (T0) in cognitive and motor assessment at an expected average of 1 week (T1), 2 months (T2) and 3 months (T3).
  Cognition and motor performance will be also measured with standardized paper and pencil tests, scales and questionnaires using the three dimensions of the International Classification of Functioning (Body structure and function / Activity limitation / Participation restriction).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lejeune, Principal Investigator — St. Luc Hospital; Gaëtan Stoquart, Principal Investigator — St. Luc Hospital; Martin Edwards, Principal Investigator — Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Centre Hospitalier Neurologique William Lennox, Ottignies, Brabant Wallon
  - Cliniques Universitaires St Luc, Woluwé-Saint-Lambert, Brussels Capital

REFERENCES:
- [Derived] Doumas I, Lejeune T, Edwards M, Stoquart G, Vandermeeren Y, Dehez B, Dehem S. Clinical validation of an individualized auto-adaptative serious game for combined cognitive and upper limb motor robotic rehabilitation after stroke. J Neuroeng Rehabil. 2025 Jan 23;22(1):10. doi: 10.1186/s12984-025-01551-w. PMID 39849588
- [Derived] Dehem S, Montedoro V, Brouwers I, Edwards MG, Detrembleur C, Stoquart G, Renders A, Heins S, Dehez B, Lejeune T. Validation of a robot serious game assessment protocol for upper limb motor impairment in children with cerebral palsy. NeuroRehabilitation. 2019;45(2):137-149. doi: 10.3233/NRE-192745. PMID 31498135
- [Derived] Montedoro V, Alsamour M, Dehem S, Lejeune T, Dehez B, Edwards MG. Robot Diagnosis Test for Egocentric and Allocentric Hemineglect. Arch Clin Neuropsychol. 2019 Jun 1;34(4):481-494. doi: 10.1093/arclin/acy062. PMID 30084880